CLINICAL TRIAL: NCT00478504
Title: Double Blind Cross-over Randomized Controlled Trial Comparing Letrozole Versus Clomifene Citrate for Ovulation Induction in Women With Polycystic Ovarian Syndrome
Brief Title: Letrozole Versus Clomifene Citrate for Ovulation Induction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Saad Amer, Associate Professor, University of Nottingham
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RD-5103-015-06; EudraCT No: 2006-006514-15
Record Dates: First submitted 2007-05-23; First posted 2007-05-24 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Infertility; Polycystic Ovarian Syndrome
Keywords: anovulation; ovulation induction,; polycystic ovarian syndrome; clomifene citrate; letrozole
MeSH Terms: conditions — Infertility; Polycystic Ovary Syndrome; Anovulation | interventions — Letrozole; Clomiphene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clomiphene citrate (Active Comparator): Starting daily dose 50 mg on menstrual cycles days 2 to 6, to be increased to 100 mg daily if there is no response to 50 mg
  Interventions: Drug: Clomifene citrate
- Letrozole (Active Comparator): Starting daily dose 2.5 mg on menstrual cycles days 2 to 6, to be increased to 5 mg daily if there is no response to 2.5 mg
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Letrozole — Starting daily dose 2.5 mg on menstrual cycles days 2 to 6, to be increased to 5 mg daily if there is no response to 2.5 mg
  Arms: Letrozole
Drug: Clomifene citrate — Starting daily dose 50 mg on menstrual cycles days 2 to 6, to be increased to 100 mg daily if there is no response to 50 mg
  Arms: Clomiphene citrate

SUMMARY:
The primary aim of the study is to assess the efficacy of letrozole as an ovulation induction agent and to test the hypothesis that letrozole will generate better pregnancy rates with fewer multiple pregnancies and higher live birth rate than the current standard agent, clomifene citrate in anovular infertile women with polycystic ovarian syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 - 39
2. BMI < 36
3. Infertility due to anovulation
4. PCOS: At least two of the following diagnostic criteria of:

   1. Oligo/amenorrhoea
   2. Hyperandrogenaemia: biochemical (testosterone ≥2.5 nmol/l or free androgen index (FAI) ≥ 5) or clinical (acne/hirsutism) evidence
   3. USS evidence of PCO (either ≥12 follicles measuring 2-9 mm in diameter, or an ovarian volume of > 10 ml)
5. No recent (within 6 months) treatment for induction of ovulation
6. Normal semen analysis (WHO 1999)
7. Proven patency of at least one Fallopian tube

Exclusion Criteria:

1. Inability to give informed consent
2. Contraindication to letrozole or clomifene citrate
3. Absence of any inclusion criteria

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 159 (Actual)
Dates: Start 2007-05; Primary Completion 2014-06 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Pregnancy rate | 14 moths

SECONDARY OUTCOMES:
1. Ovulation rate 2. Number of growing and mature follicles during treatment 3. Miscarriage rate 4. Live-birth rate 5. Multiple pregnancy rate 6. Endometrial thickness | 14 months

CONTACTS AND LOCATIONS:
Overall Officials: Saad Amer, MD, MRCOG, Principal Investigator — University of Nottingham and Derby Hospitals NHS foundation Trust
Locations (1):
- Royal Derby Hospital, Derby, Derbyshire, United Kingdom

REFERENCES:
- [Derived] Amer SA, Smith J, Mahran A, Fox P, Fakis A. Double-blind randomized controlled trial of letrozole versus clomiphene citrate in subfertile women with polycystic ovarian syndrome. Hum Reprod. 2017 Aug 1;32(8):1631-1638. doi: 10.1093/humrep/dex227. PMID 28854590
- See also: Related Info — http://www.derbyhospitals.nhs.uk/research/
- See also: Lay summary of the trial — http://saadamer.com/clet-trial-for-pcos/
- See also: Patient information sheet — http://saadamer.com/docs/CLET_Patient_information_sheet.pdf